CLINICAL TRIAL: NCT06802861
Title: Relationship Between Aspirin Metabolism and Markers of Metabolic Dysfunction Among Pregnant Persons at Risk of Pre-eclampsia
Acronym: RAMP
Status: Recruiting | Type: Observational
Sponsor: University of Tennessee Graduate School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 5316
Record Dates: First submitted 2025-01-24; First posted 2025-01-31 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-01

CONDITIONS: Preeclampsia; Preeclampsia (PE); Preeclampsia (PE) Risk; Obesity and Obesity-related Medical Conditions; Pregnancy; Pregnancy Complications; Gestational Diabetes; Gestational Diabetes Mellitus in Pregnancy; Gestational Complications
Keywords: metabolic dysfunction; gestational diabetes; pregnancy; maternal obesity; maternal insulin resistance; aspirin metabolism; GDM; substrate oxidation; gestational glucose intolerance
MeSH Terms: conditions — Pre-Eclampsia; Obesity; Pregnancy Complications; Diabetes, Gestational; Pregnancy in Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pregnant individuals at risk for preecampsia

SUMMARY:
This study's primary purpose is to determine the relationship between aspirin metabolism and markers of metabolic dysfunction among patients at risk for preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

* Recommended aspirin for pre-eclampsia prevention by OB/GYN or MFM specialist based on ACOG and USPSTF guidelines (1 high risk factor, 2+ moderate risk factors)

  * Willingness to adhere to aspirin therapy
  * Willingness to undergo 2h OGTT for serum and urine collection in addition to survey collection, indirect calorimetry, body composition measures, neonatal measures, etc.
  * Gestational age at enrollment <16 weeks
  * Ability to speak, read, and communicate via English

Exclusion Criteria:

* Type 2 Diabetes Mellitus

  * Type 1 Diabetes Mellitus
  * Current gestational diabetes mellitus
  * Current/active platelet disorder or bleeding diathesis (thrombocytopenia of any etiology, idiopathic thrombocytopenic purpura/ITP, thrombotic thrombocytopenic purpura/TTP, von Willebrand disease, etc.)
  * Thrombophilia
  * Current use of NSAID for other indication (indomethacin, ibuprofen, etc.)
  * Current use of other immune-modulating agents and biologics (hydroxychloroquine, azathioprine, 6-mercaptopurine, IL-6 inhibitors, etc.)
  * Current or recent use of steroids
  * Current use of prophylactic or therapeutic anticoagulation
  * Medical contraindication to aspirin therapy
  * Molar pregnancy
  * Renal disease
  * Inability or unwillingness to give informed consent
  * Current psychiatric illness/social situation that would limit compliance with study requirements, as determined by the principal investigators

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Limited to the biological sex of female, during pregnancy
Study Population: Pregnant individuals at risk for preeclampsia
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Hexadecadienoate (z score) | 60 minutes after ingestion of 75 grams of glucose during a single study visit between 14-20 weeks gestational age
  Hexadecadienoate (long chain poly unsaturated fatty acid metabolite obtained from metabolomics assay) (z score)
Salicylate (z score) | 60 minutes after ingestion of 75 grams of glucose during a single study visit between 14-20 weeks gestational age
  Salicylate (benzoate metabolite obtained from metabolomics assay)(z score)

SECONDARY OUTCOMES:
Urinary thromboxane B2 level (pg/mg creat) | 60 minutes after ingestion of 75 grams of glucose, during a single study visit between 14-20 weeks gestational age
  Urinary thromboxane B2 level (pg/mg creat)
Fasting Salicylate level (ug/mL) | Fasting, at the beginning of a single study visit between 14-20 weeks gestational age
  Fasting Salicylate level (ug/mL) in venous blood
1 Hour Salicylate level (ug/mL) | 60 minutes after ingestion of 75 grams of glucose during a single study visit between 14-20 weeks gestational age
  1 Hour Salicylate level (ug/mL) in venous blood
2 Hour Salicylate level (ug/mL) | 120 minutes after ingestion of 75 grams of glucose during a single study visit between 14-20 weeks gestational age
  2 Hour Salicylate level (ug/mL) in venous blood
Fasting PFA-100 epinephrine closure time | Fasting, at the beginning of a single study visit between 14-20 weeks gestational age
  Fasting PFA-100 epinephrine closure time in venous blood
1 Hour PFA-100 epinephrine closure time | 60 minutes after ingestion of 75 grams of glucose during a single study visit between 14-20 weeks gestational age
  1 Hour PFA-100 epinephrine closure time in venous blood
2 Hour PFA-100 epinephrine closure time | 120 minutes after ingestion of 75 grams of glucose during a single study visit between 14-20 weeks gestational age
  2 Hour PFA-100 epinephrine closure time in venous blood
Homeostatic Model Assessment for Insulin Resistance | Calculated from fasting insulin and fasting glucose collected at the start of a single study visit between 14-20 weeks gestational age
  Approximates insulin resistance.
Fasting Resting Metabolic Rate | Measured at the start of a single study visit between 14-20 weeks gestational age
  Resting metabolic rate describes whole body caloric expenditure, which is assessed using indirect calorimetry
Fasting Respiratory Quotient | Measured at the start of a single study visit between 14-20 weeks gestational age
  Resting respiratory quotient describes whole body caloric expenditure, which is assessed using indirect calorimetry
Fasting Carbohydrate Oxidation Rate | Measured at the start of a single study visit between 14-20 weeks gestational age
  Fasting carbohydrate oxidation rate measures whole body carbohydrate oxidation, which is assessed using indirect calorimetry
Fasting Lipid Oxidation Rate | Measured at the start of a single study visit between 14-20 weeks gestational age
  Fasting lipid oxidation rate measures whole body lipid oxidation, which is assessed using indirect calorimetry
Fasting Insulin (mIU/mL) | Fasting, at the beginning of a single study visit between 14-20 weeks gestational age
  Fasting insulin level (mIU/mL) in venous blood
Fasting glucose (mg/dL) | Fasting, at the beginning of a single study visit between 14-20 weeks gestational age
  Fasting glucose level (mg/dL) in venous blood
Fasting lactate (mmol/L) | Fasting, at the beginning of a single study visit between 14-20 weeks gestational age
  Fasting lactate level (mmol/L) in venous blood
Fasting triglycerides (mg/dL) | Fasting, at the beginning of a single study visit between 14-20 weeks gestational age
  Fasting triglycerides level (mg/dL) in venous blood
Fasting high density lipoprotein (mg/dL) | Fasting, at the beginning of a single study visit between 14-20 weeks gestational age
  Fasting high density lipoprotein level (HDL) (mg/dL) in venous blood
Fasting very low density lipoprotein (mg/dL) | Fasting, at the beginning of a single study visit between 14-20 weeks gestational age
  Fasting very low density lipoprotein level (VLDL) (mg/dL) in venous blood
Fasting low density lipoprotein (mg/dL) | Fasting, at the beginning of a single study visit between 14-20 weeks gestational age
  Fasting low density lipoprotein level (LDL) (mg/dL) in venous blood
Fasting cholesterol (mg/dL) | Fasting, at the beginning of a single study visit between 14-20 weeks gestational age
  Fasting cholesterol level (mg/dL) in venous blood
Fasting free fatty acids (mEq/L) | Fasting, at the beginning of a single study visit between 14-20 weeks gestational age
  Fasting free fatty acids (FFA) (mEq/L) in venous blood

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tennessee Medical Center, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Reasonable requests will be considered on a case-by-case basis.
Supporting Information: Study Protocol
Time Frame: We anticipate publishing the study protocol within the next 2 years